CLINICAL TRIAL: NCT06575660
Title: Digital Support for Mental Health Intervention in Patients With Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB24-0605
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Inflammatory Bowel Diseases; Anxiety; Depression; Ulcerative Colitis; Crohn Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Anxiety Disorders; Depression; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with IBD who self-report mild to moderate levels of anxiety or depression (Experimental)
  Interventions: Behavioral: Mental health support session

INTERVENTIONS:
Behavioral: Mental health support session — a single AI-VR mental health support session using the XAIA application

SUMMARY:
This is a small, exploratory study that will investigate using an artificial intelligence (AI) and virtual reality (VR), digital wellness application (app) to deliver a mental health support session in outpatient and hospitalized patients with inflammatory bowel disease (IBD) and co-existing symptoms of mild to moderate anxiety or depression.

The purpose of this study is to explore if a mental health support session using the app is feasible, safe, and acceptable to IBD patients and whether it could possibly help with physical and comorbid psychological symptoms of these patients.

DETAILED DESCRIPTION:
The mental health support session is delivered by a virtual reality digital wellness application (app). The app is a Chat GPT-4 powered AI and VR platform called XAIA (eXtended reality Artificially Intelligent Ally). [Chat GPT is an AI program that generates dialogue.] The app is publicly available on the Apple Vision Pro (a VR tool). It was developed by a group of providers, including a psychiatrist, at Cedars-Sinai Medical Center to devise a scalable solution for the increasing demand for mental wellness experiences. The application uses the combination of an AI-powered virtual avatar, named "XAIA," and a VR environment to deliver immersive and personalized mental health support in mixed-reality environments.

This is a mixed method study with primarily a qualitative focus. Patients with IBD who self-report mild to moderate levels of anxiety or depression will be invited to try a single AI-VR mental health support session using the XAIA app. Participant observations, experiences, and opinions of the application will be collected through surveys and semi-structured interviews. Pre- and post- session pain and state anxiety scores will be collected.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* Patients with Inflammatory Bowel Disease (Crohn's Disease or Ulcerative Colitis)
* English-speaking
* Patients with score of 5-14 on General Anxiety Disorder-7 (GAD-7) questionnaire or 5-19 on Patient Health Questionnaire-9 (PHQ-9) within 3 months
* Able to provide written consent

Exclusion Criteria:

* Unwilling and/or unable to participate
* Non-English speakers
* Self-reported history of severe motion sickness
* The presence of a facial/head deformity that will prohibit comfortably wearing of a VR headset
* Legally blind or deaf
* Having had a seizure in the past year
* Unable to understand the instructions or to consent to participation in the study.
* Those who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
Determine the feasibility of utilizing a GPT-4-powered AI-VR mental health support session in patients with IBD | Day 1 post-session
  Measured via a post-session, semi-structured interview
Determine the safety of utilizing a GPT-4-powered AI-VR mental health support session in patients with IBD | Day 1 post-session
  Measured by proportion of subjects with at least one adverse event
Determine the patient acceptance of utilizing a GPT-4-powered AI-VR mental health support session in patients with IBD | Day 1 post-session
  Measured via Session Rating Scale (SRS V.3.0), which is a visual analogue scale that measures self-reported effective therapeutic relationships. Scores range from 0 to 40, with higher scores indicating more effective relationships. Scores are commonly classified as "any score lower than 36 overall, or 9 on any [of the 4] scale[s], could be a source of concern..."

SECONDARY OUTCOMES:
To assess change in pain scores pre- and post-session | Day 1 pre-session; Day 1 post-session
  Measured via Visual Analogue Pain Scale, which is a scale that measures self-reported pain intensity. Scores range from 0-10, with higher scores indicating greater pain intensity. Scores are commonly classified as "no pain" (0), "mild pain" (1-3), "moderate to severe pain" (4-6), "very severe pain" (7-9), "worst possible pain" (10).
To assess change in mood scores pre- and post-session | Day 1 pre-session; Day 1 post-session
  Spielberger State-Trait Anxiety Inventory (STAI), which is a tool that measures self-reported anxiety. Scores range from 0-40, with higher scores indicating greater anxiety. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).
To characterize any limitations for creating a AI-VR mental health support tool optimally aligned with the needs of patients with IBD | Day 1 post-session
  Measured via a post-session, semi-structured interview
To characterize any potential future improvements for creating a AI-VR mental health support tool optimally aligned with the needs of patients with IBD | Day 1 post-session
  Measured via a post-session, semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: David T Rubin, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States